CLINICAL TRIAL: NCT00124540
Title: Misoprostol for Preventing Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: University of Witwatersrand, South Africa (Other); Effective Care Research Unit (Other); Family Care International (Other)
Responsible Party: Justus Hofmyer, University of Witwatersrand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2.4.5
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Postpartum Hemorrhage
Keywords: Misoprostol; Active management; Postpartum hemorrhage; Maternal morbidity; Anemia; Developing countries
MeSH Terms: conditions — Postpartum Hemorrhage; Anemia | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator): placebo resembling misoprostol
  Interventions: Drug: placebo
- 2 (Experimental): misoprostol
  Interventions: Drug: misoprostol

INTERVENTIONS:
Drug: misoprostol
  Arms: 2
Drug: placebo — placebo resembling misoprosotl
  Arms: 1

SUMMARY:
This hospital-based, multicenter, randomized, placebo-controlled trial will assess the effects of misoprostol as part of active management of the third stage of labor on postpartum blood loss, complications, and side effects. Twelve hundred eligible women will receive routine oxytocics (oxytocin 5-10 IU) plus either 400 mcg sublingual misoprostol or placebo during or immediately after delivery. The primary outcome will be measured blood loss of =>500 mls within one hour after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Women who have given birth to 1 or more live-born infants (para 1 or more)
* Vaginal delivery

Exclusion Criteria:

* Refusal or inability to give informed consent
* Delivery regarded as abortion according to local gestational age limits
* Inability to take misoprostol sublingually
* Cesarean section
* Assisted vaginal delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Blood loss =>500 mls within one hour after enrollment

SECONDARY OUTCOMES:
Blood loss =>1000 mls within one hour after enrollment
Mean blood loss after enrollment
Blood transfusion
Hemoglobin level <8 g/dL 24 hours after delivery
Maternal morbidity and mortality
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Lindeka Mangesi, Study Director — Effective Care Research Unit, East London Hospital Complex, South Africa; G. J. Hofmeyr, MD, Principal Investigator — Effective Care Research Unit, Frere Maternity Hospital, East London Hospital Complex
Locations (5):
- University College Hospital, Ibadan, Nigeria
- South Africa (3):
  - Tembisa Hospital, Johannesburg
  - Rob Ferreira Hospital, Mbombela
  - Dora Nginza Hospital, Port Elizabeth
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Hofmeyr GJ, Fawole B, Mugerwa K, Godi NP, Blignaut Q, Mangesi L, Singata M, Brady L, Blum J. Administration of 400 mug of misoprostol to augment routine active management of the third stage of labor. Int J Gynaecol Obstet. 2011 Feb;112(2):98-102. doi: 10.1016/j.ijgo.2010.08.019. Epub 2010 Dec 4. PMID 21130990